CLINICAL TRIAL: NCT06009536
Title: Does Resistance Training Protocol Change Micromorphology in Achilles Tendinopathy?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Motol (Other)
Responsible Party: Principal Investigator, Stanislav Machač, Ph.D, Academic woorker, University Hospital, Motol
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EK-402 /22b
Record Dates: First submitted 2023-08-19; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-04

CONDITIONS: Achilles Tendinopathy
Keywords: Achilles Tendinopathy; Ultrasonography; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance training protocol (Experimental): Participants in this group will complete a 12-week ankle dorsiflexion resistance training protocol according to Silbernagel. It is a series of heel rise exercises with a gradual progression of load according to defined criteria, which the patient practices every day.
  Interventions: Other: Achilles Tendon Loading Exercise Protocol According to Silbernagel
- Participants with healthy tendons (No Intervention): Participants in this group are considered healthy based on subjective judgment followed by clinical and ultrasound examination of the Achilles tendon.
  In this group, no specific treatment will be performed, only Achilles tendon will be monitored through time.

INTERVENTIONS:
Other: Achilles Tendon Loading Exercise Protocol According to Silbernagel — It is a 12-week Silbernagel ankle dorsiflexion resistance training protocol. It is a series of exercises with a gradual progression of load according to defined criteria, which the patient practices every day.
  Arms: Resistance training protocol

SUMMARY:
This work is designed as a prospective cohort study, in which the effects of a protocol of 12-week resistance training loading the Achilles tendon in patients with Achilles tendinopathy (AT) will be monitored. It is estimated that at least 20 patients will participate. In addition, there will be a small control group of healthy participants which will not complete the same protocol, but will be monitored for natural changes in same objectives. Group of patients will be instructed to perform a training protocol.

DETAILED DESCRIPTION:
The research within one participant will last a total of 26 weeks from the initial to the final examination and will include control measurements at 6 and 12 weeks from the beginning of therapy. Potential participants will be selected based on the recommendation of a specialist doctor and their suitability will be assessed according to the inclusion criteria. They will then be invited to an initial examination. This will include an objective examination by a physiotherapist, a subjective assessment by the patient and an ultrasonographic (USG) examination followed by a micromorphological analysis using special software. At the end of the initial examination, the participant will be informed about training protocol.

ELIGIBILITY:
Inclusion Criteria:

* the patient shows symptoms of Achilles tendinopathy (pain, swelling and dysfunction in the area of Achilles tendon), which at least partially limit his quality of life during normal or sporting activities,
* the patient is in the age group of 18-60 years,
* the patient has difficulties in only one lower limb; the second, asymptomatic limb will be considered the reference,
* the patient is not aware of any mechanical damage to the tendon in symptomatic limb in the past (e.g. partial or complete rupture as a result of an injury),
* the patient has not undergone any treatment aimed at AS in the last 3 months (surgery, corticoid application, plasma therapy, shock waves, physiotherapy, etc.), objective US examination of AS shows structural changes (expansion, neovascularization, focal hypoechoic areas, etc.).

Exclusion Criteria:

* patient has been diagnosed with a rheumatic disease or a disease of the central nervous system
* patient is aware of mechanical damage to the Achilles tendon as a result of an injury in the past.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in Peak Spatial Frequency Radius at the site of Pathology | Change of initial values at 26 weeks follow up after beginning of the therapy.
  Measured by spatial frequency analysis software from ultrasound picture in mm-1. In a linear view with specific settings of ultrasound machine, the site of the largest pathology is selected, then the image is saved and uploaded to the software that evaluates the PSFR parameter.
Change in Tendon Diameter at the Place of Maximum Tendon Width | Change of initial values at 26 weeks follow up after beginning of the therapy.
  Measured by tools in ultrasound machine in mm2. In linear view is selected maximal width place, then the tendon diameter is measured using device tools.

SECONDARY OUTCOMES:
Change in VISA-A Questionnaire Score | Change of initial values at 39 weeks follow up after beginning of the therapy.
  The VISA-A questionnaire is standardized questionnaire for patients with Achilles tendinopathy. The results are recorded in points (0-100 points). The higher score indicates patients better condition.

CONTACTS AND LOCATIONS:
Overall Officials: Stanislav Machac, PhD, Study Chair — University Hospital Motol and 2nd Faculty of Medicine, Charles University
Locations (1):
- University Hospital Motol and 2nd Faculty of Medicine, Charles University, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No